CLINICAL TRIAL: NCT01165931
Title: A Study to Compare the Acute Coronary Vasodilating Effects of the sGC Stimulator Riociguat (BAY 63-2521) With the Nitric Oxide Donor Nitroglycerin in Patients With Coronary Artery Disease
Brief Title: Coronary Vasomotor Response After Riociguat Exposure
Acronym: CORONARIES
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14550
Record Dates: First submitted 2010-07-15; First posted 2010-07-20 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (BAY63-2521) — 0.1 mg intracoronary infusion through coronary guide catheter. Single dose. Sequential application after initial vasoactive bolus of Adenosine (non-study drug) and Nitroglycerin (non-study drug).

SUMMARY:
The aim of the study is to assess the effects of intracoronary Riociguat on coronary blood flow in subjects with coronary artery disease and to compare this effect with the intracoronary nitroglycerin, a coronary vasodilator widly used to treat patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with coronary artery disease

Exclusion Criteria:

* Patents with coronary artery disease with >/= 70% luminal stenosis by coronary angiography in one of the 3 major epicardial coronary arteries (left anterior descending artery [LAD], left circumflex coronary artery [LCX] or right coronary artery [RCA]) undergoing cardiac catheterization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The ratio of the coronary blood flow after Riociguat to the corresponding flow observed after adenosine, compared to that after nitroglycerin administration | Within 5 min after completion of the intracoronary Riociguat infusion

SECONDARY OUTCOMES:
Adverse event collection | Until 30 days after study drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Boston, Massachusetts, United States